CLINICAL TRIAL: NCT01957748
Title: CCTG 594: Engagement and Retention in Care for HIV+, A Multicenter Trial of the California Collaborative Treatment Group
Brief Title: CCTG 594: Engagement and Retention in Care for HIV+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of California, Los Angeles (Other); University of Southern California (Other); City of Long Beach Department of Health and Human Services (Other Government); California HIV/AIDS Research Program (Other)
Responsible Party: Principal Investigator, Maile Young Karris, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CCTG 594
Record Dates: First submitted 2013-09-09; First posted 2013-10-08 (Estimated); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Patient Adherence; HIV Positive
Keywords: Retention; Care; Engagement
MeSH Terms: conditions — Patient Compliance; HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (SoC) (No Intervention): Subjects randomized to the Standard of Care Arm will receive their HIV clinic's current standard of care retention services.
- SoC + ALERT Intervention (Active Comparator): Subjects randomized into the ALERT Enhanced Retention Intervention Arm will receive SoC at the HIV clinic where subjects are seen. In addition to SoC, the Intervention arm will receive aggressive engagement efforts by the ALERT specialist to ensure visit continuity and retention into care. The ALERT specialist will also administer an education intervention consisting of 5 retention modules designed to improve HIV knowledge and self-efficacy, and will also monitor health care visits and intervene via methods to track, find, and re-engage patients during the study.
  Interventions: Behavioral: SoC + ALERT Intervention

INTERVENTIONS:
Behavioral: SoC + ALERT Intervention — Enhanced retention efforts and education modules will be implemented by the ALERT Specialist to ensure retention to care.
  Arms: SoC + ALERT Intervention

SUMMARY:
CCTG 594 is a controlled, unblinded, two-arm, randomized (1:1) clinical trial to evaluate the effectiveness of a clinic-based HIV ALERT specialist on improving endpoints of retention in care and maintenance of ART as compared to the current standard of care (SoC) in HIV primary care clinics.

DETAILED DESCRIPTION:
Design: CCTG 594 is a controlled, unblinded, two-arm, randomized (1:1) clinical trial to evaluate the effectiveness of a clinic-based HIV ALERT specialist on improving endpoints of retention in care and maintenance of ART as compared to the current standard of care (SoC) in HIV primary care clinics.

Duration: Each subject will receive follow-up of at least 48 weeks.

Sample Size: A total of 300 subjects will be randomized, 150 per arm.

Study Population: Eligible subjects will include 1) newly diagnosed HIV-infected individuals entering primary HIV care at one of the CCTG clinics, or 2) previously diagnosed HIV-infected individuals who are "out of care" defined as having no visit with a prescribing HIV provider in the last 180 days and not on a stable ARV regimen.

Stratification: Subjects will be stratified based on study site and if they are newly diagnosed or returning to care.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, as documented by any licensed screening antibody test, such as ELISA, and confirmed by a second antibody test, such as Western blot, or detectable plasma HIV-1 RNA at any time prior to study entry. If an ELISA or Western blot is not available, HIV infection may be documented by two HIV RNA values ≥2000 copies/mL, drawn at least 24 hours apart. The RNA assays must have been run at a CLIA-approved laboratory or equivalent.
* 18 years of age or older.
* Able to give written informed consent.
* New patient to the clinic (defined as someone who has never engaged in HIV care) or a patient returning to care (defined as a patient previously seen at least once by a prescribing HIV provider who has not seen a prescribing HIV provider in the last 180 days and is not on a stable ARV regimen).
* English or Spanish Speaking.
* Registered to receive HIV primary care services at one of the identified CCTG-affiliated clinic, i.e. the Owen Clinic at UC San Diego Health System, Harbor-UCLA Medical Center clinic or Rand Schrader clinic at USC.

Exclusion Criteria:

* Unstable neurologic, psychiatric, or physical condition which, in the opinion of the investigator, would limit participation with study procedures for the duration of the study.
* A level of drug or alcohol use that, in the opinion of the investigator, would preclude safe participation in the study.
* Resident of nursing home or skilled facility.
* Pregnant or breastfeeding.
* Patient's first primary care visit (for new patients) or return to care visit (for patients returning to care) occurred > 60 days ago.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2013-10-08 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Time to lost to follow up | Baseline to Week 48
  The CCTG 594 primary outcome is "time to lost to follow up." Lost to follow up is defined as "no visit with a prescribing HIV provider in the last 180 days. All randomized subjects will be followed for a minimum of 48 weeks. Subjects that do not meet the primary endpoint by the time the study ends will be censored.

SECONDARY OUTCOMES:
Time to initiation of ART | Baseline to Week 48
  The CCTG 594 secondary outcome is "time to initiation of ART." All randomized subjects will be followed for a minimum of 48 weeks. Subjects that do not initiate ART will be censored at their last visit date.

OTHER OUTCOMES:
Descriptive analyses | Baseline to two years
  Descriptive secondary analyses comparing the two randomized groups will include:
  * Baseline and follow-up scores on HIV and health literacy assessments, disclosure rates, adherence, and measures of self-efficacy
  * Number of primary care visits per year
  * HIV RNA < 50 and <200 copies/mL at years 1 and 2
  * CD4 cell counts and changes from baseline in CD4 at years 1 through 2
  * Scores on Beck Depression Index
  * Substance use
  * HIV high-risk transmission behaviors
  * Time to AIDS diagnosis or death
Return to Care after Primary Endpoint | Baseline to 2 years
  Proportions of subjects that meet the primary endpoint but subsequently return to care will be compared between the randomized groups. The times between last visit and return visit will also be compared between the randomized groups.

CONTACTS AND LOCATIONS:
Overall Officials: Maile Karris, MD, Principal Investigator — CCTG, UCSD AVRC, UCSD Owen Clinic; Katya Calvo, MD, Study Chair — CCTG, Harbor-UCLA
Locations (3):
- United States (3):
  - University Southern California, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - Harbor-UCLA Medical Center, Torrance, California

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT01957748/Prot_SAP_000.pdf